CLINICAL TRIAL: NCT00249600
Title: Lower-Cost Contingency Management in a Group Setting
Brief Title: Lower-Cost Contingency Management in a Group Setting - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-14618-1; R01DA014618 (NIH); R01-14618-1
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Substance Abuse
Keywords: contingency management; substance abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Contingency management

SUMMARY:
The purpose of this study is to evaluate the efficacy of prize contingency management (CM) in enhancing attendance, reducing drug use, and improving health among clients attending two HIV drop-in centers. Specifically, 172 clients are randomly assigned to one of two 6-month treatment conditions: standard 12-step oriented group treatment, or CM group treatment. In the CM group, clients earn the chance to win prizes for submitting clean urine specimens and for complying with steps toward their treatment goals. Activities related to improving health will be emphasized, such as attending medical appointments, recording daily medication consumption, getting prescriptions filled, and attending medication adherence support groups. Group attendance, drug use, medical problems, services received, and risky drug use and sexual behaviors will be measured pre-treatment and at months 1, 3, 6, 9 and 12.

ELIGIBILITY:
Inclusion criteria:

* HIV-positive and a member of The Living Center or the Manchester Area Network on AIDS
* DSM-IV diagnosis of current opioid or cocaine abuse or dependence
* willingness to accept random assignment to one of the two treatment groups

Exclusion criteria:

* inability to comprehend the study (Mini-mental status score <21; Folstein & Folstein, 1975; or inability to pass an informed consent quiz)
* severely disruptive behavior
* in recovery for pathological gambling (due to potential similarity between the CM procedure and gambling)
* non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2003-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Drug use | baseline and each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States